CLINICAL TRIAL: NCT05289947
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Efficacy and Safety of MLC1501 in Patients With Stroke
Brief Title: MLC1501 Study Assessing Efficacy in Post STrOke Subjects With mOtor Deficits
Acronym: MAESTOSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFSA2021_01
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Stroke, Ischemic; Strokes Thrombotic; Stroke Sequelae; Stroke, Cardiovascular; Stroke, Embolic; Stroke, Cryptogenic
Keywords: stroke; MLC1501; MAESTOSO; stroke recovery; neurorestoration
MeSH Terms: conditions — Stroke; Ischemic Stroke; Thrombotic Stroke; Myocardial Infarction; Embolic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 500-mg placebo capsule, 4 capsules twice a day for 24 weeks
  Interventions: Other: Placebo
- MLC1501 Low-dose (Active Comparator): MLC1501 low-dose 500-mg capsule, 4 capsules twice a day for 24 weeks
  Interventions: Drug: MLC1501
- MLC1501 High-dose (Active Comparator): MLC1501 high-dose 500-mg capsule, 4 capsules twice a day for 24 weeks
  Interventions: Drug: MLC1501

INTERVENTIONS:
Other: Placebo — Caramel, chocolate brown, flavor (E_1982648), dextrin
  Arms: Placebo
Drug: MLC1501 — Powdered extract of Radix astragali, Rhizoma chuanxiong, Radix angelica sinensis, Radix polygala
  Arms: MLC1501 High-dose; MLC1501 Low-dose

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled trial of MLC1501 in patients with stroke. Eligible participants will be randomized in a 1:1:1 ratio to orally receive MLC1501 high-dose twice a day, MLC1501 low-dose twice a day, or matching placebo for 24 weeks.

DETAILED DESCRIPTION:
A total of 300 patients will be included with approximately 100 patients randomized to each treatment arm. Randomization will be performed centrally and stratified according to the following factors at the time of randomization: country, National Institute of Health Stroke Scale (NIHSS) (8 to 12, 13 to 18) and received either intravenous or endovascular thrombolysis/thrombectomy (no, yes).

Efficacy clinical assessments will include Fugl-Meyer motor Assessment (FMA), modified Rankin Scale (mRS), Patient Reported outcome Measurement Information System - Global Health (PROMIS-10) and NIHSS.

Each patient will undergo standard safety assessments including physical exam and laboratory parameters, and be observed for adverse events for the duration of the study. Electrocardiogram (ECG), hematology, clinical chemistry, coagulation, and urinalysis will be performed at specified intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* ≥18 years old or legal age as per country requirement
* Diagnosed with acute ischemic stroke with compatible brain imaging findings between 2 days to 10 days (inclusive) prior to inclusion.
* NIHSS total score of 8 to 18 (inclusive) at the time of inclusion with a combined score of at least 3 on the NIHSS motor items 5A or 5B and/or 6A or 6B.
* A candidate for active rehabilitation in the opinion of the treating physician.
* Able to comply with the requirements of the protocol and provide written informed consent by patient or legal representative before any study-specific procedure is performed.

Exclusion Criteria:

* Pre-stroke modified Rankin score of >1.
* Contraindication to any of the study procedures.
* Patients who became medically unstable within 24 hours after intravenous or endovascular thrombolysis or thrombectomy.
* Intake of any herbal or traditional medicine within the past 30 days.
* Participation in another investigational drug or device trial within the past 30 days.
* Intake of warfarin in the past one week or expected to be on warfarin while in the study.
* Women who are pregnant or wish to continue breastfeeding while in the study. Women of child-bearing potential may be included if they agree to strict abstinence or use of effective contraception, except systemically acting hormonal contraceptives. Hormone replacement therapy in menopausal/post-menopausal or surgically sterilized women is also not allowed while in the study.
* Any known food allergy or hypersensitivity to Astragalus membranaceus, Ligusticum chuanxiong, Polygala tenuifolia, Angelica sinensis, or members of the Fabaceae/Leguminosae family (e.g., legume, pea, bean), Polygalaceae family (e.g., milkwort, snakeroot), Apiaceae/Umbelliferae family (e.g., anise, caraway, carrot, celery, dill, parsley, parsnip), or Quillaja bark (soapbark).
* Evidence of other significant non-ischemic brain lesion which could affect long-term function or disability.
* Evidence of advanced medical condition that would affect study assessment and follow-up, such as cancer, renal failure, liver cirrhosis, severe dementia, or psychosis.
* Any other medical or psychiatric or cognitive condition which, in the study investigator's opinion, may jeopardize the patient by his/her participation in this study, may hamper his/her ability to complete procedures required in the study, affect study assessment and follow-up, or affect the validity of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer motor Assessment (FMA) | 24 weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia

SECONDARY OUTCOMES:
Adverse events | up to 24 weeks
  Listing and calculating the number and percentage of subjects experiencing non-serious and serious adverse events for each dose cohort
Fugl-Meyer motor Assessment (FMA) | 12 and 24 weeks
modified Rankin Scale (mRS) | 4, 12 and 24 weeks
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 (no symptoms at all) to 5 (severe disability). A separate category of 6 is usually added for patients who expire.
Patient Reported Outcome Measurement Information System - Global Health (PROMIS-10) | 4, 12 and 24 weeks
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
National Institute of Health Stroke Scale (NIHSS) | 12 and 24 weeks
  The maximum possible score is 42 (severe), with the minimum score being a 0 (no symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chen, BMBCh, MRCP, FAMS, FRCPE, Principal Investigator — Departments of Pharmacology and Psychological Medicine, National University of Singapore
Locations (11):
- Philippines (7):
  - Metro Davao Medical And Research Center, Davao City, Davao Region
  - Quirino Memorial Medical Center, Manila, Manila
  - University of Santo Tomas Hospital, Manila, Manila
  - Baguio General Hospital and Medical Center, Baguio City
  - West Visayas State University Medical Center, Iloilo City
  - Jose R. Reyes Memorial Medical Center, Manila
  - Manila Doctors Hospita, Manila
- Singapore (4):
  - Changi General Hospital, Singapore, Singapore
  - National Neuroscience Institute (NNI) @ Tan Tock Seng Hospital (TTSH), Singapore, Singapore
  - Raffles Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Once decided, only anonymized IPD may be shared with other collaborative stroke trials consortiums.

REFERENCES:
- [Derived] Chen CPLH, Esagunde RU, Escabillas CG, Hiyadan JH, Advincula JM, Co COC, Collantes MEV, Lao AY, Koh YH, De Silva DA, Tham CH, Lokin JK, Venketasubramanian N. Phase II randomised, double-blind, placebo-controlled trial to assess the efficacy and safety of MLC1501 in patients with stroke: the MLC1501 study Assessing Efficacy in post-STrOke Subjects with mOtor deficits (MAESTOSO) study protocol. Stroke Vasc Neurol. 2025 Oct 27;10(5):657-664. doi: 10.1136/svn-2024-003750. PMID 39915229